CLINICAL TRIAL: NCT01228838
Title: A Multicenter Randomized, Double-Blind, Controlled Study to Evaluate Safety, Tolerability and Preliminary Efficacy of Two Capsaicin Concentration Variations of NGX-1998 (10% or 20% w/w) in Subjects With Postherpetic Neuralgia (PHN)
Brief Title: Study of NGX-1998 for the Treatment of Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurogesX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C204
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2011-05

CONDITIONS: Postherpetic Neuralgia; Pain
Keywords: postherpetic neuralgia; PHN; capsaicin; herpes zoster; shingles; analgesics; neuropathy
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain; Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NGX-1998, 10% w/w capsaicin (Experimental)
  Interventions: Drug: NGX-1998
- NGX-1998, 20% w/w capsaicin (Experimental)
  Interventions: Drug: NGX-1998
- Placebo liquid (Placebo Comparator)
  Interventions: Drug: Placebo Liquid

INTERVENTIONS:
Drug: NGX-1998 — Capsaicin topical liquid to be applied for 5 minutes one time only.
  Arms: NGX-1998, 10% w/w capsaicin; NGX-1998, 20% w/w capsaicin
Drug: Placebo Liquid — Placebo topical liquid to be applied for 5 minutes one time only.
  Arms: Placebo liquid

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of NGX-1998 applied for 5 minutes for the treatment of postherpetic neuralgia (PHN).

DETAILED DESCRIPTION:
This study is a 12-week multicenter randomized, double-blind, controlled evaluation of the efficacy, safety and tolerability of NGX-1998 for the treatment of postherpetic neuralgia (PHN). Eligible subjects will have pain from PHN, with average numeric pain rating scale (NPRS) scores during screening of 4 to 9 (inclusive). Painful areas of up to 1500 cm2 will be treated during a single Test Article application. Subjects will be randomly assigned to receive NGX-1998 (10% or 20% w/w) or placebo according to an unequal allocation scheme of 2:2:1. Subjects will also be stratified by gender.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 90 years of age, inclusive.
* Diagnosis of PHN with at least six (6) months of pain since shingles vesicle crusting.
* Average NPRS scores for PHN-associated pain during Days -14 to -4 of 4 to 9, inclusive.
* Intact, unbroken skin over the painful area(s) to be treated.
* If taking chronic pain medications, be on a stable (not PRN) regimen for at least 21 days prior to Test Article Application Visit and willing to maintain medications at same stable dose(s) and schedule throughout the study.
* Female subjects with child-bearing potential must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test, to be performed within 7 days of the Test Article Application Visit.
* All subjects must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study.
* If breastfeeding, the subject should agree not to breastfeed their child after treatment on the treatment day.
* Be willing and able to comply with protocol requirements for the duration of study participation.
* Subjects must sign an informed consent form for this study approved by the Investigator's Institutional Review Board/Independent Ethics Committee (IRB/IEC).

Exclusion Criteria:

* Concomitant opioid medication, unless orally or transdermally administered and not exceeding a total daily dose of morphine 60 mg/day, or equivalent. Parenteral opioid use is excluded.
* Unavailability of an effective medication for treatment related discomfort for the subject, such as unwillingness to use opioid analgesics during study treatment, or high tolerance to opioids precluding the ability to relieve treatment-associated discomfort.
* Active substance abuse or history of chronic substance abuse within the past year, or prior chronic substance abuse judged likely to recur during the study period.
* Recent use (within 21 days preceding the Test Article Application Visit [Day 0]) of any topically applied pain medication on the painful areas.
* Receipt of Qutenza® within 12 months of the Test Article Application Visit (Day 0). Subjects who have received Qutenza® 12 months or more before Test Article Application Visit (Day 0), and who did not respond should also be excluded.
* Participation in another drug research study within 30 days preceding the Test Article Application Visit (Day 0).
* Current use of any Class I anti-arrhythmic drugs or III anti-arrhythmic drugs.
* Diabetes mellitus, unless well-controlled as evidenced by an HBA1c level less than or equal to nine percent (9%).
* A recent history of cardiovascular or cerebrovascular events or unstable hypertension, unless adequately controlled by medication.
* Significant pain of an etiology other than PHN, for example, compression-related neuropathies, fibromyalgia or arthritis.
* Painful PHN areas located on the face, above the hairline of the scalp, and/or in proximity to mucous membranes.
* Any implanted medical device for the treatment of neuropathic pain.
* History of hypersensitivity to capsaicin, local anesthetics or any components of the CTLs, Cleansing Gel or the lidocaine (2.5%) / prilocaine (2.5%) topical anesthetic cream.
* Patients with glucose-6 phosphate dehydrogenase deficiencies.
* Significant ongoing or untreated abnormalities or conditions, including active malignancy defined as treatment required in the last five (5) years, that in the opinion of the Investigator would interfere with the ability to complete the study or the evaluation of AEs.
* Patients with congenital or idiopathic methemoglobinemia.
* Recent history of a significant medical-surgical intervention in the judgment of the Investigator; examples include but are not limited to major surgery or percutaneous angioplasty/coronary artery stent placement within the past 3 months, and receipt of immunosuppressive therapy within 3 months, prior to the Test Article Application Visit [Day 0].
* Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete daily pain diaries requiring subject's recall of average PHN pain level in the past 24 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in the "average pain for the past 24 hours" NPRS score during Weeks 2-8. | Weeks 2-8

SECONDARY OUTCOMES:
Absolute change and percent change from baseline in the "average pain for the past 24 hours" NPRS score at Week 8 and 12 | Week 8 and Week 12
Absolute change and percent change from baseline in the "average pain for the past 24 hours" NPRS score during Weeks 2-12. | Weeks 2-12
Proportion of subjects with at least a 30% decrease from baseline in their "average pain for the past 24 hours" NPRS during Weeks 2-8, Weeks 2-12, at Week 8 and Week 12. | Weeks 2-12
Proportion of subjects with at least a 2 unit decrease from baseline in their "average pain for the past 24 hours" NPRS during Weeks 2-8, Weeks 2-12, at Week 8 and Week 12. | Week 8 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Trudy Vanhove, MD, PhD, MBA, Study Director — NeurogesX
Locations (35):
- United States (35):
  - NeurogesX Investigational Site, Huntsville, Alabama
  - NeurogesX Investigational Site, Tucson, Arizona
  - NeurogesX Investigational Site, Irvine, California
  - NeurogesX Investigational Site, La Jolla, California
  - NeurogesX Investigational Site, Napa, California
  - NeurogesX Investigational Site, San Francisco, California
  - NeurogesX Investigational Site, Santa Monica, California
  - NeurogesX Investigational Site, New Port Richey, Florida
  - NeurogesX Investigational Site, North Palm Beach, Florida
  - NeurogesX Investigational Site, Sarasota, Florida
  - NeurogesX Investigational Site, St. Petersburg, Florida
  - NeurogesX Investigational Site, Marietta, Georgia
  - NeurogesX Investigational Site, Boise, Idaho
  - NeurogesX Investigational Site, Bloomington, Illinois
  - NeurogesX Investigational Site, West Des Moines, Iowa
  - NeurogesX Investigational Site, Kansas City, Kansas
  - NeurogesX Investigational Site, Lexington, Kentucky
  - NeurogesX Investigational Site, Shreveport, Louisiana
  - NeurogesX Investigational Site, Hyannis, Massachusetts
  - NeurogesX Investigational Site, Ann Arbor, Michigan
  - NeurogesX Investigational Site, Minneapolis, Minnesota
  - NeurogesX Investigational Site, Hattiesburg, Mississippi
  - NeurogesX Investigational Site, Albany, New York
  - NeurogesX Investigational Site, Rochester, New York
  - NeurogesX Investigational Site, Hickory, North Carolina
  - NeurogesX Investigational Site, Winston-Salem, North Carolina
  - NeurogesX Investigational Site, Portland, Oregon
  - NeurogesX Investigational Site, Altoona, Pennsylvania
  - NeurogesX Investigational Site, San Antonio, Texas
  - NeurogesX Investigational Site, Webster, Texas
  - NeurogesX Investigational Site, Salt Lake City, Utah
  - NeurogesX Investigational Site, Richmond, Virginia
  - NeurogesX Investigational Site, Seattle, Washington
  - NeurogesX Investigational Site, Wenatchee, Washington
  - NeurogesX Investigational Site, Madison, Wisconsin